CLINICAL TRIAL: NCT02847338
Title: Comparison of Optimal Hypertension Regimens (Part of the Ancestry Informative Markers in Hypertension (AIMHY) Programme - AIMHY-INFORM)
Brief Title: Comparison of Optimal Hypertension Regimens
Acronym: AIMHY-INFORM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Dr Ian B Wilkinson, Consultant, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AO94005
Record Dates: First submitted 2016-06-30; First posted 2016-07-28 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Lisinopril; Amiloride; Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mono-therapy group (Experimental): The monotherapy group will be treated with the following treatments:
  A) 1 to 2 weeks of Amlodipine 5mg followed by 6 to 7 weeks of Amlodipine 10mg B) 1 to 2 weeks of Lisinopril 10mg followed by 6 to 7 weeks of Lisinopril 20mg C) Approximately 8 weeks of 25mg Chlortalidone
  Participants will be randomly allocated to one of six possible sequences of treatments of the three-treatment-three period Williams design: ABC, ACB, BAC, BCA, CAB, and CBA.
  Interventions: Drug: Amlodipine; Drug: Lisinopril; Drug: Chlortalidone
- Dual-therapy arm (Experimental): The dual-therapy group will be treated with the following treatments:
  A) Approximately 8 weeks of Amlodipine 5mg and Lisinopril 20mg B) Approximately 8 weeks of Amlodipine 5mg and Chlortalidone 25mg C) Approximately 8 weeks of Lisinopril 20mg and Chlortalidone 25mg D) Approximately 8 weeks of Amiloride 10mg and Chlortalidone 25mg
  Participants will be randomly allocated to one of four possible sequences of treatments of the four-treatment four-period Williams design: ABDC, BCAD, CDBA, and DACB.
  Interventions: Drug: Amlodipine; Drug: Lisinopril; Drug: Amiloride; Drug: Chlortalidone

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 5mg and Amlodipine 10mg will be one of the treatments in which patients will receive on the monotherapy arm and on the dual therapy arm.
Drug: Lisinopril — Lisinopril 10mg and Lisinopril 20mg will be one of the treatments in which patients will receive on the monotherapy arm.
  Lisinopril 20mg will be one of the treatments in which patients will receive on the dual therapy arm.
Drug: Amiloride — Amiloride 10mg will be one of the treatments in which patients will receive on the dual therapy arm.
  Arms: Dual-therapy arm
Drug: Chlortalidone — Chlortalidone 25mg will be one of the treatments in which patients will receive on the dual therapy arm and monotherapy arm.

SUMMARY:
High blood pressure (Hypertension) is extremely common and is a major cause of heart disease, kidney disease and stroke. One in three of the UK (United Kingdom) population will require treatment for hypertension at some point in their lives. A healthy lifestyle alone is often not enough to control blood pressure, and drug treatment is usually required. Although a wide variety of drugs are available to treat hypertension, choosing the right kind of tablet or combination of tablets for individual patients is a problem, and therefore many people have poor blood pressure control.

Hypertension treatment within the UK is currently selected according to age and self-defined ethnicity (SDE). There are limitations to this approach which include wide variability in the response to hypertension drug classes between people. There is also uncertainty about selecting hypertension drugs for ethnic minorities other than those of African/Caribbean ancestry, for example, South Asians because of a lack of information from trials. In the AIM HY-INFORM study the investigators are looking to recruit equal number of black/caribbean, south asian and white european participants to be able to compare differences in hypertension treatments and ethnicity.

The primary objective of this study is to determine if the response to antihypertensive drugs differs by self defined ethnicity.

DETAILED DESCRIPTION:
In the UK, current NICE (National Institute for Health and Clinical Excellence) guidance stratifies hypertension treatment according to age and self-defined ethnicity (SDE). Different initial monotherapies are recommended for all those aged over 55 years, and for younger black compared to white individuals. However, there is no recommended stratification for combination therapy. The evidence based supporting the current guidance on SDE stratification is limited, and there is a specific lack of data from UK based populations.

Stratification based on SDE has a number of limitations and an alternative approach is stratification based on ancestry informative markers (AIM). There are genetic polymorphisms, which show substantially different frequencies between populations from different geographical regions, and can predict geographical ancestry with remarkable accuracy. AIM are thus more likely to capture the genetic component of variation in drug response in ethnically diverse population.

Metabolomic profiling of plasma and urine may provide complementary information to AIM, as differences between individuals will reflect both genetic and environmental influences. To address these issues the investigators intend to compare the variation in response to antihypertensive drug treatments in three SDE cohorts, and relate this to variation in AIM and metabolomic profiles. Our objective is to test the validity of current NICE guidance on antihypertensives stratification based on SDE, to provide evidence about SDE stratification for dual therapy, and to examine whether more effective personalisation of antihypertensive treatment, can be achieved using AIM and/or metabolomic profiling.

An assessment of patient stratification based on AIM phenotypes against SDE will enable the selection of optimal and more effective choices of anti-hypertensive treatments from currently existing first line drugs (and combinations of) and ultimately reduce the attrition of antihypertensive therapies.

Output from the trial will provide the first perspective evidence for best treatment choice according to SDE for white, black and asian populations in the UK. This should reduce the number of consultations; time required to achieve optimal blood pressure control and the contribution to between hypertension control in the UK.

Patients in the trial will be enrolled on a monotherapy or dual therapy regime depending on their history of hypertension. The monotherapy group of patients will enter a randomised, open-label, three-treatment three-period cross over trial.

The dual therapy group of patients will enter a randomised, open-label, four-treatment four-period cross over trial.

Randomisation, for each crossover design, will be stratified by three SDE groups.

The duration for individual participants will be approximately 24 (monotherapy) or 32 weeks (dual therapy)

The hypertensive medication used in this trial are:

Amlodipine 5 or 10mg, Chlortalidone 25mg, Amiloride 10mg, Lisinopril 10 or 20mg,

Participants on the dual therapy treatment arm will have a total of 11 visits including screening/enrolment (visit 1) and baseline visit (visit 2)

Participants on the monotherapy treatment arm will have a total of 9 visits including screening/enrolment (visit 1) and baseline visit (visit 2)

A total number of 1320 participants will be enrolled in the study across participating sites, so that approximately 660 participants in each therapy regime (approximately 220 participants per ethnic group) complete the trial.

An optional skin-sodium investigation will be conducted at selected sites only where capacity and capability to complete the sub study investigations is demonstrated. The sub study aims to recruit up to 60 participants who have already given consent for the main AIM HY INFORM Trial. Consent for the optional sub-study will be obtained separately.

The investigation comprises two optional assessments: a skin biopsy and a sodium magnetic resonance imaging (23Na MRI) scan. Both assessments will be used to quantify skin sodium levels. Participants in the mono and dual therapy arms can elect to have the skin biopsy, the MRI scan, or both, at the baseline visit. Participants in the mono therapy arm only, can elect to have the skin biopsy, the MRI scan, or both, following completion of the amlodipine (A) and chlortalidone (C) study arms. The additional measurements are not anticipated to take more than approximately 2 hours.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial the participant must:

1. Have given written informed consent to participate
2. Be aged 18 to 65 years inclusive
3. Self-Define Ethnicity: participants should SELF IDENTIFY into 1 of the three groups below:

   White White British White Irish Any other white background

   Black or Black British Black Caribbean Black African Any other black background

   Asian or Asian British Asian Indian Asian Pakistani Asian Bangladeshi Any other Asian background
4. Be hypertensive defined as:- Mono-therapy rotation

   1. currently untreated with EITHER an ABPM day time average blood pressure ≥ 135mmHG (systolic) or ≥ 85mmHg (diastolic) OR Home BP measurements using a validated device based on the average of 10 blood pressure readings of ≥135 mmHg (systolic) or ≥85 mmHg (diastolic)
   2. Patients who may be taking antihypertensive drugs at sub therapeutic doses or in ineffective combinations, and who are felt likely to be controllable on a study drug and willing and able to be washed out, at the discretion of the CI (Chief Investigator) / PI (Principal Investigator), can enter the trial if they meet the above criteria.

Dual therapy rotation

a.Treated hypertensive receiving one to three antihypertensive drugs with a blood pressure (ABPM daytime average blood pressure or Home BP as in a.) between 135 or 200 mmHg (systolic) AND between 85 or 110 mmHg (diastolic).

Exclusion Criteria:

The presence of any of the following will mean participants are ineligible:

* Participant does not fit into one of the defined ethnic groups e.g. Mixed
* Pregnant or breastfeeding women
* Known or suspected secondary hypertension
* Significant sensitivity or contraindications to any of the study medications
* Participants taking lithium or are regularly consuming non-steroidal anti-inflammatory drugs at variable doses
* Requirement to take any of the study drugs continuously e.g. ACEi and heart failure
* Any clinically significant hepatic impairment
* Any clinically significant kidney impairment
* Concurrent participation in another clinical trial using systemic vasoactive medications or medications known to interact with the study drugs (participation in another study as part of the AIM HY mechanistic or social science programme will not be an exclusion criterion)
* Patients who are deemed unsuitable by the investigator on clinical grounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Actual)
Dates: Start 2016-11; Primary Completion 2023-10 (Actual); Study Completion 2023-10 (Actual)

PRIMARY OUTCOMES:
Seated Automated Office Systolic Blood Pressure | Approximately 8 weeks after receiving each treatment up to week 24 for mono therapy patients and up to week 32 for dual therapy patients
  This is planned for all participants

SECONDARY OUTCOMES:
Seated Automatic office systolic blood pressure | At every visit - every 4 weeks up to week 24 for mono therapy patients and every 4 weeks up to week 32 for dual therapy patients. From screening until last visit.
  This is planned for all participants
Core Cardiovascular Measurements | Core cardiovascular measurements will be performed on all participants at Baseline. For all patients there is an option for them to have the measurements repeated at weeks 8, 16, 24 Mono&Dual and week 32 Dual only, these subsequent visits are optional.
  This is planned for all participants, but is only mandatory at baseline
Detailed Self Defined Ethnicity | Screening visit only
  This is planned for all participants
Ambulatory Blood Pressure and/or blood pressure | This will be measured for a subgroup of patients at Baseline, week 8, week 16, week 24 Dual&Mono & week 32 Dual only
  This is planned for a subgroup of patients who agree to participate in the sub-study
Optional Cardiovascular measures | These measurements will be performed on a subgroup of patients at Baseline, week 8, week 16, week 24 Dual&Mono & week 32 Dual only
  This is planned for a subgroup of patients who agree to participate in the sub-study

OTHER OUTCOMES:
Baseline demographic comparison | Baseline visit
  This is planned for all participants
Urine compliance drug screen | These will be measured for a subgroup of patients at Baseline visit, week 8, week 16, week 24 Dual&Mono & week 32 Dual only
  This is planned for a random subgroup of participants who are taking part in the sub-study

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wilkinson, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (14):
- United Kingdom (14):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - Queen Elizabeth Hospital, Birmingham
  - Sandwell & West Birmingham Hospitals NHS Trust, Birmingham
  - Heartlands Hospital, Birmingham
  - University Hospital Llandough, Cardiff
  - University of Glasgow, Glasgow
  - Liverpool Heart and Chest Hospital, Liverpool
  - William Harvey Research Institute, Barts and the London Medical School, London
  - St Thomas' Hospital, London
  - St George's Hospital, London
  - Hammersmith & Fulham GP Partnership: Richford Gate Medical Practice, London
  - Manchester Royal Infirmary, Manchester
  - Nottingham University Hospital: QMC Campus, Nottingham
  - Lister Hospital, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Only after the investigator has finished with the data and not patient identifiable data

REFERENCES:
- [Derived] Wych J, Grayling MJ, Mander AP. Sample size re-estimation in crossover trials: application to the AIM HY-INFORM study. Trials. 2019 Dec 2;20(1):665. doi: 10.1186/s13063-019-3724-6. PMID 31791376
- [Derived] Mukhtar O, Cheriyan J, Cockcroft JR, Collier D, Coulson JM, Dasgupta I, Faconti L, Glover M, Heagerty AM, Khong TK, Lip GYH, Mander AP, Marchong MN, Martin U, McDonnell BJ, McEniery CM, Padmanabhan S, Saxena M, Sever PJ, Shiel JI, Wych J, Chowienczyk PJ, Wilkinson IB. A randomized controlled crossover trial evaluating differential responses to antihypertensive drugs (used as mono- or dual therapy) on the basis of ethnicity: The comparIsoN oF Optimal Hypertension RegiMens; part of the Ancestry Informative Markers in HYpertension program-AIM-HY INFORM trial. Am Heart J. 2018 Oct;204:102-108. doi: 10.1016/j.ahj.2018.05.006. Epub 2018 May 20. PMID 30092411